CLINICAL TRIAL: NCT01465750
Title: Epidemiology of Ovarian Cancer in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201103108RC
Record Dates: First submitted 2011-10-26; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovarian Cancer

SUMMARY:
Cancer is the leading cause of mortality in the investigators country. According to the statistics of the Department of Health, the incidence of ovarian cancer increased in recent years and the mortality rate is highest in all gynecologic malignancies in Taiwan. Ovarian cancer becomes a more and more important disease gradually in the field of gynecologic malignancies. The classification of histology in ovarian cancer included epithelial ovarian cancer、germ cell tumors、sex-cord cell tumors…etc. Epithelial ovarian carcinoma is the most common ovarian cancer clinically. Early diagnosis is difficult due to the lack of obvious initial symptoms, so ovarian cancer patients are usually at advanced stage when the diagnosis is confirmed. The prognostic parameters for ovarian carcinomas include tumor stage, histological subtype, degree of malignancy, residual tumor after surgical intervention and the response to chemotherapy. However, the possible etiology and mechanism of ovarian cancer is still unclear. However, there is no epidemiologic data of ovarian cancer in Taiwan. Therefore the investigators propose this study to use Taiwan registry database provided by Department of Health to analyze the epidemiology and prognosis of ovarian cancer patients in Taiwan.

DETAILED DESCRIPTION:
Study population: To evaluate the epidemiology and prognosis of ovarian cancer in Taiwan, we will conduct a nationwide analysis through linking national cancer registry database. Every citizen in Taiwan has a life-long identification number to link individual information, including health status. The Taiwan household registry database provided by Department of Health will be the source population. National household registry and death certificate will be adopted to ascertain the live status of study subjects, and provided individual demographic characteristics.All individual linkages between databases will be conducted according to the study protocols, i.e. databases will be linked by corresponding identification number, name (Chinese characters) and birthday, and all data included in this study will be analyzed without individual identification information. The agreement of utilizing the databases in the study was obtained from the Bureau of Health Promotion in Taiwan.

Incident and death cases ascertainment: Patients with ovarian cancer, including epithelial ovarian carcinoma, germ cell tumors, sex cord tumors … etc., will be identified from computerized linkage to the Taiwan national cancer registry with International Classification of Diseases for Oncology Third Edition T-code C569. Histological types will be identified from morphology code in the cancer registry database. Women affected by ovarian cancer and found death due to ovarian cancer (International Classification of Diseases 9th edition code 183) in deaths certificate will be defined as death cases.

Statistical Analyses: The numbers of person-years at risk of developing and dying for ovarian cancer will be calculated. Incidence rates will be calculated by dividing the number of ovarian cancer cases by the person-years at risk of developing ovarian cancer. Mortality rates will be calculated by dividing the number of ovarian cancer deaths by the person-years at risk of dying from ovarian cancer. The association between mortality and age, histology, time periods will be estimated through Kaplan-Meier survival analysis and Cox's proportional hazards model. It is defined as significantly different statistically when p value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients of ovarian cancer registered at National Taiwan Cancer registration system between 1979-2008

Exclusion Criteria:

nil

Ages: 15 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ovarian cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From diagnosis of ovarian cancer to death or last date of linked data available from the Taiwan Cancer Registry or Death Certification Profile
  The follow-up of each participant (in personyears) was calculated from the date of enrollment to the date of ovarian cancer diagnosis, date of death, or last date of linked data available from the Taiwan Cancer Registry or Death Certification Profile, whichever came first until December 31, 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan